CLINICAL TRIAL: NCT03902275
Title: Validation of a Quantra Supported Hemotherapy Algorithm in Cardiac Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: SARS-CoV-2 Pandemic
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: HemoSonics LLC (Industry)
Responsible Party: Principal Investigator, Dr. med. Florian Raimann, Principal investigator, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 42/19
Record Dates: First submitted 2019-03-26; First posted 2019-04-04 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Hemorrhage; Bleeding
Keywords: cardiac surgery; bleeding; point of care testing; POCT; algorithm based therapy
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quantra (Experimental): Evaluation of bloodsamples using the Quantra and Multiplate device
  Interventions: Other: Quantra-Algorithm
- Control (Active Comparator): Evaluation of bloodsamples using the ROTEM and Multiplate device
  Interventions: Other: ROTEM-Algorithm

INTERVENTIONS:
Other: Quantra-Algorithm — Hemotherapy based on Quantra-Algorithm
  Arms: Quantra
Other: ROTEM-Algorithm — Hemotherapy based on Basic-Algorithm
  Arms: Control

SUMMARY:
The aim of this study is to develop a coagulation algorithm based on Quantra POCT for the treatment of coagulopathic cardiac surgery patients.

DETAILED DESCRIPTION:
In order to perform a targeted coagulation therapy during intra- and postoperative care of cardiosurgical patients, it is necessary to know the hemostatic potential. After blood samples have been taken for coagulation diagnosis, they are usually sent to the central laboratory. After analysis and validation, the results are transmitted electronically. The loss of time due to sample transport, analysis and provision of the results prolongs the time required to derive therapeutic measures.

In recent years, point of care testing (POCT) devices for the diagnosis of coagulopathic patients have become increasingly important. In our clinic, POCT devices have been routinely used for intra- and postoperative targeted coagulation therapy for years. These include the ROTEM delta and Multiplate. For analysis, a whole blood sample is pipetted together with test reagents. Depending on the selected reagent, different parts of the coagulation cascade can be evaluated and, depending on this, an appropriate therapy can be derived. A coagulation algorithm developed in our clinic is based on these measurement results and has been used successfully for years for perioperative coagulation management. This algorithm requires additional information on the platelet function, which is also carried out as standard on the bed side using multi-plate analysis as POCT.

A new system for whole blood analysis has recently become available on the market. The Quantra from HemoSonics also allows the analysis of a whole blood sample on the bed side. Due to the cassette structure, the time-consuming and potentially error-prone pipetting of a whole blood sample is no longer necessary. The aim of this study is to develop a coagulation algorithm based on Quantra POCT for the treatment of coagulopathic cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

>18 years elective operation with cardiac bypass

Exclusion Criteria:

participation on another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Bloodloss | From finishing operation until 24 hours postoperative
  Cumulative bloodloss directly after surgery for 24h Determined by cumulative volume of all drains in millilitres

SECONDARY OUTCOMES:
Correlations of parameters between POCT and laboratory parameters. | During operation within 24 hours postoperative
  Quick
Correlations of parameters between POCT and laboratory parameters. | During operation within 24 hours postoperative
  prothrombine time
Correlations of parameters between POCT and laboratory parameters. | During operation within 24 hours postoperative
  activated partial thromboplastin time
Correlations of parameters between POCT and laboratory parameters. | During operation within 24 hours postoperative
  Firbinogen
Correlations of parameters between POCT and laboratory parameters. | During operation within 24h postoperative
  platelet count
Multiplate results | During operation within 24 hours postoperative
  Determin platelet function with TRAP test
Multiplate results | During operation within 24 hours postoperative
  Determin platelet function with ASPI test
Multiplate results | During operation within 24 hours postoperative
  Determin platelet function with ADP test
Time saving by using a cassette | During operation within 24 hours postoperative
  Influence of a cassette structure in comparison to pipetting with regard to the temporal availability of the measurement results
Use of blood products | During operation within 24 hours postoperative
  Cumulative volume of administered fresh frozen plasma, platelet infusion and packed red blood cells in mililitres
Coagulationfactos and procoagulant drugs | During operation within 24 hours postoperative
  Cumulative usage of prothrombin complexe concentrate measured in international units, fibrinogen measured in gramm, tranexamic acid measured in gramm, desmopressin measured in microgramm, Calcium measured in gramm, activated factor VII measured in international units
Thromboembolic complications | During operation within 24h postoperative
  Thromboembolic complications
Comorbidities | 15 years before operation
  Comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Florian J Raimann, Dr. med., Principal Investigator — Goethe University
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weber CF, Zacharowski K, Brun K, Volk T, Martin EO, Hofer S, Kreuer S. [Basic algorithm for Point-of-Care based hemotherapy: perioperative treatment of coagulopathic patients]. Anaesthesist. 2013 Jun;62(6):464-72. doi: 10.1007/s00101-013-2184-8. German. PMID 23793973
- [Result] Ferrante EA, Blasier KR, Givens TB, Lloyd CA, Fischer TJ, Viola F. A Novel Device for the Evaluation of Hemostatic Function in Critical Care Settings. Anesth Analg. 2016 Dec;123(6):1372-1379. doi: 10.1213/ANE.0000000000001413. PMID 27224934
- [Result] Viola F, Lin-Schmidt X, Bhamidipati C, Haverstick DM, Walker WF, Ailawadi G, Lawrence MB. Sonorheometry assessment of platelet function in cardiopulmonary bypass patients: Correlation of blood clot stiffness with platelet integrin alphaIIbbeta3 activity, aspirin usage, and transfusion risk. Thromb Res. 2016 Feb;138:96-102. doi: 10.1016/j.thromres.2015.11.036. Epub 2015 Nov 26. PMID 26688324
- [Result] Huffmyer JL, Fernandez LG, Haghighian C, Terkawi AS, Groves DS. Comparison of SEER Sonorheometry With Rotational Thromboelastometry and Laboratory Parameters in Cardiac Surgery. Anesth Analg. 2016 Dec;123(6):1390-1399. doi: 10.1213/ANE.0000000000001507. PMID 27749339
- [Result] Reynolds PS, Middleton P, McCarthy H, Spiess BD. A Comparison of a New Ultrasound-Based Whole Blood Viscoelastic Test (SEER Sonorheometry) Versus Thromboelastography in Cardiac Surgery. Anesth Analg. 2016 Dec;123(6):1400-1407. doi: 10.1213/ANE.0000000000001362. PMID 27159065
- [Derived] Michel S, Piekarski F, Fischer JH, Hettler V, Adam EH, Holzer L, Lotz G, Walther T, Zacharowski K, Raimann FJ. Hemostatis Analyzer-Supported Hemotherapy Algorithm in Cardiac Surgery: Protocol for a Randomized Controlled Monocentric Trial. JMIR Res Protoc. 2020 Apr 21;9(4):e17206. doi: 10.2196/17206. PMID 32314972